CLINICAL TRIAL: NCT01711294
Title: A Multicenter, Prospective, Randomized Study on Endosonographic Evaluation of Pancreatic Cystic Lesions Using 22 G, 19 G, and Flexible 19 G Fine Needle Aspiration
Brief Title: Evaluation of PCLs Using Three EUS-FNA Needles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 90869947; E7084 (Other: Boston Scientific)
Record Dates: First submitted 2012-09-26; First posted 2012-10-22 (Estimated); Results first posted 2020-11-12 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Pancreatic Cystic Lesions
Keywords: Pancreatic Cystic Lesions; PCL; EUS-FNA
MeSH Terms: interventions — Needles

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 19 G Flex Needle (Active Comparator): Device: Expect™ Endoscopic Ultrasound Aspiration Needle (19 G Flex)
  Interventions: Device: 19 G Flex Needle
- 22 G Needle (Active Comparator): Device: Expect™ Endoscopic Ultrasound Aspiration Needle (22 G)
  Interventions: Device: 22 G Needle
- 19 G Needle (Active Comparator): Device: Expect™ Endoscopic Ultrasound Aspiration Needle (19 G)
  Interventions: Device: 19 G Needle

INTERVENTIONS:
Device: 19 G Flex Needle — Fine Needle Aspiration of PCL with a 19 G Flex needle. If unsuccessful, a salvage procedure will be done with 19 G or 22 G needle.
  Arms: 19 G Flex Needle
Device: 22 G Needle — Fine Needle Aspiration of PCL with a 22 G needle. If unsuccessful, a salvage procedure will be done with 19 G Flex needle.
  Arms: 22 G Needle
Device: 19 G Needle — Fine Needle Aspiration of PCL with a 19 G needle. If unsuccessful, a salvage procedure will be done with 19 G Flex needle.
  Arms: 19 G Needle

SUMMARY:
To document impact of EUS-FNA needle size and flexibility on effectiveness of pancreatic cystic lesions (PCL) aspiration, on ability to obtain sufficient material for standard diagnostic testing, and on diagnostic accuracy of EUS-FNA aspirate for differentiation of mucinous (pre-malignant) and non-mucinous cysts.

ELIGIBILITY:
Inclusion Criteria:

* Pancreatic cystic lesion measuring 13mm or greater in largest diameter.
* Indicated for EUS evaluation of the PCL including EUS-FNA.
* Age 18 years of age or older.
* Willing and able to comply with the study procedures and provide written informed consent form to participate in the study.

Exclusion Criteria:

* Cysts in which FNA is not indicated based on review by the clinician, including potential concern of blood vessel location relative to the cyst.
* Requirement for anticoagulation using clopidogril, warfarin, or other long acting antiplatelet agents (with the exception of aspirin) that cannot be safely stopped according to institutional guidelines.
* Standard contraindications for EUS.
* Known pancreatic pseudocyst.
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2013-01-08 (Actual); Primary Completion 2017-06-06 (Actual); Study Completion 2019-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Wallace, MD,MPH, Principal Investigator — Mayo Clinic
Locations (8):
- United States (6):
  - Mayo Clinic, Scottsdale, Arizona
  - Mayo Clinic, Jacksonville, Florida
  - Indiana University Medical Center, Indianapolis, Indiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - New York Presbyterian Hospital/Columbia University Medical Center, New York, New York
- Changhai Hospital, Shanghai, China
- Asian Institute of Gastroenterology, Hyderabad, India

REFERENCES:
- [Derived] Al-Haddad M, Wallace MB, Brugge W, Lakhtakia S, Li ZS, Sethi A, Pleskow D, Nguyen CC, Pannala R, DeWitt J, Raimondo M, Woodward TA, Ramchandani MJ, Jin Z, Xu C, Faigel DO. Fine-needle aspiration of pancreatic cystic lesions: a randomized study with long-term follow-up comparing standard and flexible needles. Endoscopy. 2021 Nov;53(11):1132-1140. doi: 10.1055/a-1311-9927. Epub 2021 Feb 4. PMID 33197941

RESULTS

PARTICIPANT FLOW:
Groups:
- 19G Flex Needle: Device: Expect™ Endoscopic Ultrasound Aspiration Needle (19G Flex)
  19G Flex Needle: Fine Needle Aspiration of PCL with a 19G Flex needle. If unsuccessful, a salvage procedure will be done with 19G or 22G needle.
- 22G Needle: Device: Expect™ Endoscopic Ultrasound Aspiration Needle (22G)
  22G Needle: Fine Needle Aspiration of PCL with a 22G needle. If unsuccessful, a salvage procedure will be done with 19G Flex needle.
- 19G Needle: Device: Expect™ Endoscopic Ultrasound Aspiration Needle (19G)
  19G Needle: Fine Needle Aspiration of PCL with a 19G needle. If unsuccessful, a salvage procedure will be done with 19G Flex needle.
Period: Overall Study
Arm/Group | 19G Flex Needle | 22G Needle | 19G Needle
Started | 121 | 65 | 64
Completed | 121 | 65 | 64
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 19G Flex Needle | 22G Needle | 19G Needle | Total
Number analyzed (Participants) | 121 | 65 | 64 | 250
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (14) | 65 (16) | 62 (15) | 63 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 36 | 34 | 134
  Male | 57 | 29 | 30 | 116
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Medical History [Count of Participants; unit: Participants]
  Diabetes Mellitus | 25 | 13 | 12 | 50
  Chronic Pancreatitis | 8 | 5 | 3 | 16
  Necrotizing Pancreatitis | 0 | 1 | 0 | 1
  Symptomatic | 41 | 28 | 21 | 90
Pancreatic Cystic Lesion (PCL) Location [Count of Participants; unit: Participants]
  Head/uncinate | 53 | 30 | 26 | 109
  Body | 26 | 23 | 21 | 70
  Tail | 39 | 12 | 13 | 64
  Neck | 2 | 0 | 4 | 6
  Junction of body and tail | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Volume of Aspirated Cyst Fluid as a Function of Estimated Maximal Volume
Description: Volume of aspirated cyst fluid as a function of estimated maximal volume, based on pre-aspiration EUS measure of cyst diameter (s) (% aspiration of total estimated volume)
Time Frame: At procedure (Up to 1 hour)
Measure: Mean (Standard Deviation); unit: percentage of cyst volume aspirated
Arm/Group | 19G Flex Needle | 22G Needle | 19G Needle
Number analyzed (Participants) | 121 | 65 | 64
percentage of cyst volume aspirated | 78 (35) | 74 (39) | 73 (41)
Statistical Analysis 1: Comparison: 19G Flex Needle vs 22G Needle vs 19G Needle; Study hypothesizes that aspiration % in the 19G Flex and 19G arms would be superior by at least 10% to 22G arm, and aspiration success rate of 19G Flex would be at least 16% greater than 22G and 19G arms. Sample size calculation was performed based on the above hypotheses reached by a consensus of all collaborators and adjusted a priori; Test type: Superiority — Sample sizes were calculated using two-sample t-test for the primary endpoint and z-test for the secondary endpoint with power of 80% and two-sided alpha of 0.05. Hochberg step up procedure was used to adjust for multiple comparison. A p-value < 0.05 was considered statistically significant; p = 0.84, Wilcoxon (Mann-Whitney) — Hochberg step up procedure was used to adjust for multiple comparison; Wilcoxon was used instead of t-test because the data was not normally distributed

2. Secondary Outcome: Number of Patients With Related Adverse Events
Description: Adverse events related to study procedure or study device were tabulated. Adverse events were assessed from the index procedure up to 30 days post procedure.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | 19G Flex Needle | 22G Needle | 19G Needle
Number analyzed (Participants) | 121 | 65 | 64
Participants | 3 | 2 | 1

3. Secondary Outcome: Change in Volume of Cyst Post Initial Procedure Compared to Pre Procedure
Description: Change value is calculated as cyst volume measured after initial procedure (up to 1 hour) minus volume measured at the beginning of the initial procedure. Volume is measured using the standard geometric formula 4/3 πr³ where r is half the long axis. The volume unit is cc.
Time Frame: Procedure (Up to 1 hour)
Measure: Mean (Standard Deviation); unit: cc
Arm/Group | 19G Flex Needle | 22G Needle | 19G Needle
Number analyzed (Participants) | 121 | 65 | 64
cc | 16 (38) | 13 (35) | 22 (79)

4. Secondary Outcome: Number of Participants With Successful Echoendoscopic Fine Needle Aspiration of PCL
Description: Successful echoendoscopic fine needle aspiration of PCL, defined as complete cyst aspiration (final cyst maximal diameter of less than 5mm) or collection of aspirate adequate to perform two standard assays: cytology and carcinoembryonic antigen (CEA) (sample volume of 3 cc or more)
Time Frame: Procedure (up to 1 hour)
Measure: Count of Participants; unit: Participants
Arm/Group | 19G Flex Needle | 22G Needle | 19G Needle
Number analyzed (Participants) | 121 | 65 | 64
Participants | 108 | 53 | 48

5. Secondary Outcome: Number of Participants With PCL Reached/Penetrated
Description: Patients whose pancreatic cyst lesion(s) can be reached and penetrated by the EUS-FNA needles.
Time Frame: Procedure (Up to 1 hour)
Measure: Count of Participants; unit: Participants
Arm/Group | 19G Flex Needle | 22G Needle | 19G Needle
Number analyzed (Participants) | 121 | 65 | 64
Participants | 114 | 62 | 53

6. Secondary Outcome: Number of EUS-FNA Needle Passes at Initial Procedure.
Description: Needle pass defined as needle insertion through needle removal outside the cyst lumen, but not including needle repositioning within a single or multi-compartment cyst.
Time Frame: Procedure (Up to 1 hour)
Measure: Mean (Standard Deviation); unit: Needle passes
Arm/Group | 19G Flex Needle | 22G Needle | 19G Needle
Number analyzed (Participants) | 121 | 65 | 64
Needle passes | 1 (0) | 1 (0) | 1 (0)

7. Secondary Outcome: Number of EUS-FNA Needles Used at Initial Procedure.
Description: Total number of EUS-FNA needles used across all participants at the initial procedure.
Time Frame: Procedure (Up to 1 hour)
Measure: Number; unit: Needles used
Arm/Group | 19G Flex Needle | 22G Needle | 19G Needle
Number analyzed (Participants) | 121 | 65 | 64
Needles used | 156 | 81 | 78

8. Secondary Outcome: Time Needed for Aspiration for Each Needle Pass at Initial Procedure.
Description: Needle pass is defined as needle insertion through needle removal outside the cyst lumen, but not including needle repositioning within a single or multi-compartment cyst.
  Time of needle pass in is time of the first needle puncture into the cyst lumen. Needle pass out is time of removal of needle outside the cyst lumen, or after 10 seconds of failed attempt to aspirate fluid after the last needle re-repositioning in a single or multi-compartment cyst.
Time Frame: Procedure (Up to 1 hour)
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | 19G Flex Needle | 22G Needle | 19G Needle
Number analyzed (Participants) | 121 | 65 | 64
seconds | 86 (115) | 145 (188) | 106 (163)

9. Secondary Outcome: Time From First Needle Pass in to Last Needle Pass Out at Initial Procedure.
Description: Needle pass is defined as needle insertion through needle removal outside the cyst lumen, but not including needle repositioning within a single or multi-compartment cyst. Time of first needle pass in is time of the first needle puncture into the cyst lumen. Time of last needle pass out is time of removal of needle outside the cyst lumen at the end of the last fluid aspiration from a single or multi-loculated cyst, or after 10 seconds of failed attempt to aspirate fluid after the last needle re-repositioning in a single or multi-compartment cyst.
Time Frame: Procedure (Up to 1 hour)
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | 19G Flex Needle | 22G Needle | 19G Needle
Number analyzed (Participants) | 121 | 65 | 64
seconds | 210 (225) | 198 (161) | 238 (205)

10. Secondary Outcome: Number of Needles With Needle Insertion Rated as Excellent/Very Good
Description: Number of needles rated either Excellent or Very good when inserted into the echoendoscope at the initial procedure.
Time Frame: Procedure (Up to 1 hour)
Population: Ease of needle passage into the echoendoscope is evaluated per needle.
Measure: Count of Units; unit: Needles
Units Other Than Participants: Needles
Arm/Group | 19G Flex Needle | 22G Needle | 19G Needle
Number analyzed (Participants) | 121 | 65 | 64
Number analyzed (Needles) | 137 | 72 | 70
Needles | 89 | 65 | 31

11. Secondary Outcome: Number of Needles With Needle Removal Rated as Excellent/Very Good
Description: Number of needles rated either Excellent or Very good when removed from the echoendoscope at the initial procedure.
Time Frame: Procedure (Up to 1 hour)
Population: Ease of needle passage out of the echoendoscope is evaluated per needle.
Measure: Count of Units; unit: Needles
Units Other Than Participants: Needles
Arm/Group | 19G Flex Needle | 22G Needle | 19G Needle
Number analyzed (Participants) | 121 | 65 | 64
Number analyzed (Needles) | 135 | 72 | 70
Needles | 108 | 67 | 47

12. Secondary Outcome: Number of Needles With Needle Visualization Rated as Excellent/Very Good
Description: Number of needles rated either Excellent or Very good for visualization at the initial procedure.
Time Frame: Procedure (Up to 1 hour)
Population: Quality of needle visualization inside the cyst is evaluated per needle.
Measure: Count of Units; unit: Needle
Units Other Than Participants: Needle
Arm/Group | 19G Flex Needle | 22G Needle | 19G Needle
Number analyzed (Participants) | 121 | 65 | 64
Number analyzed (Needle) | 131 | 69 | 64
Needle | 98 | 61 | 50

13. Secondary Outcome: Number of Participants With Accurate Diagnosis of the Disease State Using the EUS-FNA Needles
Description: In order to assess the accuracy of EUS-FNA-based standard assays (cytology and CEA) as a diagnostic measure of disease state, the Disease State per EUS-FNA measure was compared to a reference diagnosis. The reference diagnostic standard was diagnosis from a surgical specimen histology, the true gold standard for cases that evolved to surgical resection within the follow-up of the study. For cases that did not progress to surgery within the follow-up period, the reference diagnostic standard was a composite diagnosis by a consensus board. The consensus board consisted of 3 experts who were blinded to the type of needle used. The consensus board diagnoses of disease state were based on baseline medical history, EUS and cross sectional imaging of the cyst, and aspirate characteristics (i.e. aspirate color and viscosity). If the EUS-FNA diagnosis matches with the histopathology or consensus board diagnosis, then the participant will be counted as having accurate diagnosis.
Time Frame: up to 2 years
Population: 3 patients excluded from analysis population in 19G Flex Arm due to histology diagnosis of neuroendocrine tumor (1), EUS diagnosis of neuroendocrine tumor (1), and solid cystic papillary neoplasm (1). 2 patients excluded from analysis population in 22G Arm due to missing EUS diagnosis (1) and EUS diagnosis of SPEN (1). 4 patients excluded from analysis population in 19G Arm due to missing EUS diagnosis (1) and EUS diagnosis of neuroendocrine tumor (3).
Measure: Count of Participants; unit: Participants
Arm/Group | 19G Flex Needle | 22G Needle | 19G Needle
Number analyzed (Participants) | 118 | 63 | 60
Participants | 91 | 50 | 50

14. Secondary Outcome: Number of Participants Requiring Post EUS-FNA Patient Management
Description: Post EUS-FNA patient management required (clinical and/or imaging surveillance, percutaneous drainage, surgical removal).
Time Frame: 30 days
Population: 3 patients excluded from this analysis (1 patient in each Arm) due to missing data in post EUS-FNA patient management.
Measure: Count of Participants; unit: Participants
Arm/Group | 19G Flex Needle | 22G Needle | 19G Needle
Number analyzed (Participants) | 120 | 64 | 63
Participants | 85 | 45 | 41

15. Secondary Outcome: Number of Participants Whose Management Decision Was Directly Influenced by the EUS Findings
Description: Patients whose Post EUS-FNA Management (clinical and/or imaging surveillance, percutaneous drainage, surgical removal) was Directly Influenced by the EUS-FNA findings.
Time Frame: Procedure - 30 days after procedure
Population: 3 patients excluded from this analysis (1 patient in each Arm) due to missing data in patient management decision directly influenced by the EUS findings.
Measure: Count of Participants; unit: Participants
Arm/Group | 19G Flex Needle | 22G Needle | 19G Needle
Number analyzed (Participants) | 120 | 64 | 63
Participants | 106 | 56 | 55

16. Secondary Outcome: Rate of Cross-over to Salvage Arm
Description: In the case of inability to access the pancreatic cystic lesion or to attain complete cyst aspiration, salvage aspiration procedure should be performed. Patients randomized to 19G Flex should undergo a salvage procedure with 22G or 19G needle (needle choice at discretion of physician); patients randomized to 22G or 19G should undergo salvage procedure with 19G Flex needle.
Time Frame: Procedure (Immediate)
Measure: Count of Participants; unit: Participants
Arm/Group | 19G Flex Needle | 22G Needle | 19G Needle
Number analyzed (Participants) | 121 | 65 | 64
Participants | 8 | 8 | 11

ADVERSE EVENTS:
Time Frame: Adverse event data collected from the time the participant signed to informed consent and was randomized to the study, until completion of the post-EUS FNA procedure 30-day follow-up visit (window of 25-35 days post EUS FNA procedure).
Description: Reported on all Serious Adverse Events and procedure-related non-serious Adverse Events.
Arm/Group | 19G Flex Needle | 22G Needle | 19G Needle
All-Cause Mortality (participants affected / at risk) | 1/121 | 1/65 | 0/64
Serious Adverse Events (participants affected / at risk) | 3/121 | 2/65 | 0/64
Other Adverse Events (participants affected / at risk) | 1/121 | 1/65 | 1/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 19G Flex Needle (N=121) | 22G Needle (N=65) | 19G Needle (N=64)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Endometrial cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Neuroendocrine carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 19G Flex Needle (N=121) | 22G Needle (N=65) | 19G Needle (N=64)
Haemorrhagic cyst (General disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2016-08-12): https://cdn.clinicaltrials.gov/large-docs/94/NCT01711294/Prot_000.pdf
  • Statistical Analysis Plan (2012-07-31): https://cdn.clinicaltrials.gov/large-docs/94/NCT01711294/SAP_001.pdf